CLINICAL TRIAL: NCT01810432
Title: Effect of Food on the Pharmacokinetics of Evacetrapib (LY2484595) in Healthy Subjects
Brief Title: Study of Food on Evacetrapib (LY2484595) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14626; I1V-MC-EIAX (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib (Fasted) (Experimental): 130 milligram (mg) oral dose of evacetrapib once daily in a fasted state for 10 days.
  Interventions: Drug: Evacetrapib
- Evacetrapib (Fed) (Experimental): 130 mg oral dose of evacetrapib once daily following a high-fat breakfast for 10 days.
  Interventions: Drug: Evacetrapib; Other: High-fat Meal

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
Other: High-fat Meal — Administered orally, at breakfast.
  Arms: Evacetrapib (Fed)

SUMMARY:
The purpose of this study is to measure how much of the drug gets into the blood stream and how long it takes the body to get rid of it when given to healthy participants. Information about any side effects that may occur will also be collected.

The study has 2 periods. In each period, participants will take the study drug for 10 days, either with or without a meal. There is a minimum 14-day washout between each period.

This study is approximately 50 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by medical history and physical examination
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m²)
* Are able to eat a high fat breakfast and abide by the food restrictions throughout the study

Exclusion Criteria:

* Have known allergies to evacetrapib, related compounds or any components of the formulation
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Are participants who currently smoke cigarettes or use tobacco or nicotine substitutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (Fast/Fed): Participants received a 130 milligram (mg) oral tablet of evacetrapib once daily (QD) for 10 days (Period 1) in a fasted state. Following a 14-day washout period participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 2) following a high-fat breakfast.
- Sequence 2 (Fed/Fasted): Participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 1) following a high-fat breakfast. Following a 14-day washout period participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 2) in a fasted state.
Period: Period 1
Arm/Group | Sequence 1 (Fast/Fed) | Sequence 2 (Fed/Fasted)
Started | 20 | 20
Received at Least 1 Dose of Study Drug | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout
Arm/Group | Sequence 1 (Fast/Fed) | Sequence 2 (Fed/Fasted)
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | Sequence 1 (Fast/Fed) | Sequence 2 (Fed/Fasted)
Started | 19 | 19
Received at Least 1 Dose of Study Drug | 19 | 19
Completed | 15 | 17
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Evacetrapib: Sequence 1-participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 1) in a fasted state. Following a 14-day washout period, participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 2) following a high-fat breakfast.
  Sequence 2-participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 1) following a high-fat breakfast. Following a 14-day washout period participants received a 130 mg oral tablet of evacetrapib QD for 10 days (Period 2) in a fasted state.
Arm/Group | Evacetrapib
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Evacetrapib
Time Frame: Day 10 Periods 1 and 2: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: All participants with evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Evacetrapib (Fasted): Participants received a 130 mg oral tablet of evacetrapib QD in a fasted state for 10 days.
- Evacetrapib (Fed): Participants received a 130 mg oral tablet of evacetrapib QD following a high-fat breakfast for 10 days.
Arm/Group | Evacetrapib (Fasted) | Evacetrapib (Fed)
Number analyzed (Participants) | 39 | 37
nanograms/milliliter (ng/mL) | 1140 (73) | 1720 (22)

2. Primary Outcome: PK: Area Under Concentration Versus Time Curve Over the 24-hour Dosing Interval (AUCτ) of Evacetrapib
Time Frame: Day 10 Periods 1 and 2: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: All participants with evaluable AUCτ data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Evacetrapib (Fasted) | Evacetrapib (Fed)
Number analyzed (Participants) | 39 | 36
nanograms*hour/milliliter (ng*h/mL) | 9930 (49) | 14400 (19)

3. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Evacetrapib
Time Frame: Day 10 Periods 1 and 2: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: All participants with evaluable tmax data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Evacetrapib (Fasted) | Evacetrapib (Fed)
Number analyzed (Participants) | 39 | 37
hours (h) | 3.00 [1.00 to 6.03] | 3.00 [1.00 to 6.00]

ADVERSE EVENTS:
Description: The total number of participants at risk in the Fasted and Fed groups is the number of participants who started Period 1 and Period 2.
Groups:
- Evacetrapib (Fasted): Participants received 130-mg oral tablet fo evacetrapib QD in a fasted state for 10 days.
- Evacetrapib (Fed): Participants received 130-mg oral tablet of evacetrapib QD following a high-fat breakfast for 10 days.
Arm/Group | Evacetrapib (Fasted) | Evacetrapib (Fed)
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 7/39 | 4/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (Fasted) (N=39) | Evacetrapib (Fed) (N=39)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.